CLINICAL TRIAL: NCT05388071
Title: The Tele-senior EMS Physician as a Strategy for the Future of Disaster Medicine - a Study Testing the Feasibility of Telemedicine in Civil Defense: Feasibility of Telemedicine Under Ambulance Station Conditions
Brief Title: Feasibility of Telemedicine Under Ambulance Station Conditions
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Anna Müller, Principal Investigator, Master of Science, Scientific Staff, RWTH Aachen University
Other Study IDs: 22-130; Notice No. 03/2019 (Other: BBK Germany)
Record Dates: First submitted 2022-05-11; First posted 2022-05-24 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Telemedicine; Disaster Medicine; Emergency Medicine
Keywords: TeleSAN; Telemedicine; Remote Consultation; Remote Treatment; Emergency Medical Services; Disaster Medicine; Emergency Medicine; Teleconsultation; Tele-emergency physician; Quality of Health Care
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention: Treatment with the aid of telemedicine: Telemedicine will be used to treat patients at an ambulance station. The medical interventions will be performed by a TeleSAN after delegation through a tele-EMS-physician if possible.
  Interventions: Other: Usage of telemedicine and tele-consultation for treatment
- No intervention: Usual treatment: Treatment will be performed as usual without the usage of telemedicine.

INTERVENTIONS:
Other: Usage of telemedicine and tele-consultation for treatment — Telemedicine will be used to treat patients at an ambulance station. The medical interventions will be performed by a TeleSAN after delegation through a tele-EMS-physician if possible.
  Groups: Intervention: Treatment with the aid of telemedicine

SUMMARY:
Our aim is to evaluate the feasibility of telemedicine in context of medical service in an ambulance station and in a further step in context of civil defense situations.

The conditions in those situations are different to the usual usage of telemedicine in context of emergency medical services (EMS) like the "Telenotarzt" in Aachen. The medical personnel who are performing the medical treatment in ambulance stations or civil defense situations are most volunteers and are ordinarily not as experienced and educated as professional medical personnel in EMS. In case of civil defense situations, the personnel also must deal with shortage in material which we are not going to simulate in our study.

The study will be realized at each one ambulance station at four large-scale events. Every time there will be a telemedicine workspace with an EMS-physician educated in telemedicine who can be contacted by briefed and equipped medical personnel according to the "TeleSAN"-standard. The emergency personnel start the patient's treatment according to their known standards and decide on their own whether they want to contact the tele-EMS-physician or not.

Before starting the tele-consultation, every patient must declare his consent to the tele-consultation, otherwise tele-consultation cannot be realized, and the patient needs to be treated according to common standards.

Due to spatial proximity of the telemedicine workspace and the ambulance station, the tele-EMS-physician can also work as an EMS-physician in the ambulance station if necessary.

As a hypothesis we declare that telemedicine is feasible in context of an ambulance station. To evaluate the feasibility, we use patient's medical protocols, observations and surveys.

DETAILED DESCRIPTION:
To evaluate the feasibility of telemedicine in context of an ambulance station with all the given restrictions compared to usage of telemedicine in emergency medical services (EMS), we will set up each one ambulance station at four large-scale events in Germany with a telemedicine infrastructure. The ambulance stations at such events are the primary place to go for visitors to get a primary medical care and is also used as a primary place for the patients of medical service providers on feet.

As part of the telemedicine infrastructure, educated personnel is required. The study protocol defines that any medical personnel with the ability to use telemedicine must be declared as a "Rettungssanitäter/in", a special paramedic qualification in Germany comparable to an EMT-I/85 (Intermediate) in the USA. These emergency personnel are called "TeleSAN".

Before the assignment in the ambulance station starts, every TeleSAN will be educated and briefed in the usage of the telemedical devices. The used equipment has been evaluated in context of the research project "TeleSAN" at the AcuteCare InnovationHub, University Hospital Aachen, Germany and is composed of a smartphone with a TeleSAN-app, a headset, and a camera. In addition to that, every TeleSAN in the ambulance station will be equipped with a Bluetooth-medical-device-set consisting of a mini-ECG, a blood glucose meter, a blood pressure cuff and a bluetooth-stethoscope which can stream all data in real-time to the tele-EMS-physician.

To stream the data and as a communication platform, the "TeleDoc"-App for video-consultation and the "TeleSAN"-App which is based on the "TeleDoc"-App with a focus on disaster medicine, both developed by Docs in Clouds TeleCare GmbH, Aachen, Germany, will be used.

Every patient who enters the ambulance station will be informed that a telemedicine-study is going on. In addition to that, the protocol defines a separate enlightenment for every patient who will be treated by telemedicine through the TeleSAN-operator before the teleconsultation starts.

Whether telemedicine will be used for patient's treatment or not is at the discretion of the TeleSAN, who will always start the treatment on his / her own and evaluates if the patient meets any exclusion criteria which would lead to not-usage of telemedicine.

In case of a none-given consent or in case of medical or technical necessity of termination of the teleconsultation, the tele-EMS-physician can work as a regular EMS-physician in the ambulance station thanks to spatial proximity. Therefore, we can guarantee a treatment according to the current medical standards all the time. In addition to the already listed medical devices, we will also have a defibrillator/ECG-monitor, a ventilator and a suction pump available for emergency situations.

The aim is to evaluate if telemedicine is feasible in context of an ambulance station regarding medical protocols, observations, and surveys.

In a further step an assessment of a possible usage of telemedicine in context of civil defense situations will be done.

ELIGIBILITY:
Inclusion Criteria:

* full legal age
* capacity to consent

Exclusion Criteria:

* apnea
* acute failure of breathing
* cardiac arrest
* STEMI
* unconsciousness
* status epilepticus
* life-threatening arrhythmia
* polytrauma
* non-manageable symptoms of a mental illness, self-endangerment, danger to others
* imminent birth
* serious traffic accident or traffic accident with children involved
* fall from a great height (>3m)
* gunshot or knife wounds to the head, neck or torso
* fire with personal damage
* high-voltage accident
* water accidents (drowning, swimming accidents, breaking in the ice)
* accidents with involvement of hazardous substances
* killing spree, hostage situations or other situations which endanger the lives of the medical personnel
* imminent threat of suizide
* non-consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We assume a cohort out of the total of festival visitors which is composed of 16-40 years old people with occasional older visitors. The patient-collective can be composed of intoxications by alcohol or drugs and minor violations of the extremities. Effects of heat and light can occur as well.
  Only those who consent to our study can be part of it, therefore every patient has to give his or her consent to the evaluation of the already bespoken outcome measures and data acquisition.
Sampling Method: Non-Probability Sample
Enrollment: 404 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-07-03 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Change of triage category using the German PRIOR algorithm (Primäres Ranking zur initialen Orientierung im Rettungsdienst) | through study completion, in total estimated 1 year
  Changes of the patient's medical condition will be measured using the german PRIOR algorithm which is used to triage patients in three categories: red, yellow and green. A change of triage category from red to yellow/green or from yellow to green means a better outcome, a change from green to yellow/red means a worse outcome.
Improvement of vital signs | through study completion, in total estimated 1 year
  Changes of the patient's medical condition will be measured by analyzing changes in the patient's vital signs. Changes from unphysiological to physiological vital signs mean a better outcome.
Improvement of NACA-Score (National Advisory Committee for Aeronautics) | through study completion, in total estimated 1 years
  Changes of the patient's medical condition will be measured using the NACA-Score. Changes from a lower to a higher score means a worse outcome.

SECONDARY OUTCOMES:
Usability of the telemedicine-devices and infrastructure and their reliable function | through study completion, in total estimated 1 year
  By analyzation of observation protocols, patient-surveys and personnel-surveys, the usability and the reliability can be evaluated

OTHER OUTCOMES:
Time for treatment | through study completion, in total estimated 1 year
  time needed for treatment using telemedicine, also regarding binding time for the physician and end of telemedicinal delegated treatment
Experience and education | through study completion, in total estimated 1 year
  Using surveys for the medical personnel, experience and education can be evaluated on the one hand for medical experience and education and on the other hand for experience an education concerning telemedicine
Acceptance of telemedicine | through study completion, in total estimated 1 year
  By analyzation of surveys an evaluation of the personnel's acceptance of telemedicine will be performed
Reasons for the usage of telemedicine | through study completion, in total estimated 1 year
  By analyzation of the medical protocols and in addition surveys and observation protocols, an evaluation of the reasons for the usage of telemedicine will be performed
Sense of security of the patients treated by teleconsultation | through study completion, in total estimated 1 year
  By analyzation of surveys and observation protocols, an evaluation of the sense of security of the patients treated by teleconsultation will be performed
Measures in the context of mass gathering medicine that can be delegated telemedically | retrospectively after all protocols have been evaluated, estimated until September 2023
  By analyzing all mission logs, the measures carried out by telemedicine and those carried out by on-site personnel without telemedicine are recorded. Subsequently, a three-stage Delphi process is carried out in which experienced tele-EMS-physicians use case descriptions to decide whether the measure can be delegated via telemedicine in the context of this case description.
Number of missions in the Accident Assistance Center that can be handled using telemedicine | retrospectively after all protocols have been evaluated, estimated until September 2023
  The results of the Delphi process (described in Outcome 10) can be used to evaluate what proportion of all cases that occurred could have been handled using telemedicine.

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Rossaint, Prof. Dr., Study Chair — University Hospital RWTH Aachen, Germany, Anaesthesiology Clinic
Locations (1):
- University Hospital RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: project page with additional information presented for lay people — https://telesan.de